CLINICAL TRIAL: NCT01964937
Title: A Phase 1b Clinical Trial to Evaluate the Safety and Immunogenicity of Different Combinations of DNAHIV-PT123, NYVAC-HIV-PT1 and NYVAC-HIV-PT4, and AIDSVAX® B/E in Healthy, HIV Uninfected Adult Participants
Brief Title: Evaluating the Safety and Immune Response to Five Different Combinations of HIV Vaccines in Healthy, HIV-Uninfected Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: IPPOX Foundation (Other); EuroVacc Foundation (Other); Global Solutions for Infectious Diseases (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 102; 11937 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX B-E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1 (Experimental): At Months 0 and 1, participants in Group 1 will receive one injection of AIDSVAX B/E ® administered intramuscularly (IM) in the right deltoid and two injections of placebo vaccine administered IM in the left deltoid.
  At Months 3 and 6, participants will receive two injections of NYVAC vaccine (NYVAC-HIV-PT1 and NYVAC-HIV-PT4) administered IM in the left deltoid and one injection of placebo vaccine administered IM in the right deltoid.
  Interventions: Biological: NYVAC-HIV-PT1; Biological: NYVAC-HIV-PT4; Biological: AIDSVAX B/E®
- Group 2 (Experimental): At Months 0 and 1, participants in Group 2 will receive two injections of NYVAC vaccine (NYVAC-HIV-PT1 and NYVAC-HIV-PT4) administered IM in the left deltoid and one injection of placebo vaccine administered IM in the right deltoid.
  At Months 3 and 6, participants will receive the AIDSVAX ® B/E vaccine administered IM in the right deltoid and two injections of placebo vaccine administered IM in the left deltoid.
  Interventions: Biological: NYVAC-HIV-PT1; Biological: NYVAC-HIV-PT4; Biological: AIDSVAX B/E®
- Group 3 (Experimental): At Months 0 and 1, participants in Group 3 will one injection of the AIDSVAX B/E vaccine administered IM in the right deltoid and one injection of placebo vaccine administered IM the left deltoid.
  At Months 3 and 6, participants will receive one injection of the DNA-HIV-PT123 vaccine administered IM in the left deltoid and one injection of placebo vaccine administered IM in the right deltoid.
  Interventions: Biological: DNA-HIV-PT123; Biological: AIDSVAX B/E®; Biological: Placebo vaccine
- Group 4 (Experimental): At Months 0 and 1, participants in Group 4 will receive one injection of the DNA-HIV-PT123 vaccine administered IM in the left deltoid and one injection of placebo vaccine administered IM in the right deltoid.
  At Months 3 and 6, participants will receive one injection of the AIDSVAX B/E ® vaccine administered IM in the right deltoid and one injection of placebo vaccine administered IM the left deltoid.
  Interventions: Biological: DNA-HIV-PT123; Biological: AIDSVAX B/E®; Biological: Placebo vaccine
- Group 5 (Experimental): At Months 0, 1, 3, and 6, participants in Group 5 will receive one injection of the DNA-HIV-PT123 vaccine administered in the left deltoid and one injection of the AIDSVAX B/E ® vaccine administered IM in the right deltoid.
  Interventions: Biological: DNA-HIV-PT123; Biological: AIDSVAX B/E®

INTERVENTIONS:
Biological: DNA-HIV-PT123 — The DNA-HIV-PT123 (containing clade C ZM96 gag and gp140 along with CN54 pol-nef) will be administered at a dose of 4 mg IM.
  Arms: Group 3; Group 4; Group 5
Biological: NYVAC-HIV-PT1 — The NYVAC-HIV-PT1 vaccine (containing clade C ZM96 gp140) will be administered at a dose of greater than or equal to 5×10^6 plaque-forming units (PFU)IM, for a planned maximum dose of 1.2×10^8 PFU.
  Arms: Group 1; Group 2
Biological: NYVAC-HIV-PT4 — The NYVAC-HIV-PT4 vaccine (containing ZM96 gag-CN54 pol-nef) will be administered at a dose of greater than or equal to 5×10^6 PFU IM, for a planned maximum dose of 1.1×10^7 PFU.
  Arms: Group 1; Group 2
Biological: AIDSVAX B/E® — The AIDSVAX B/E ® vaccine will be administered as a 1 mL/600 mcg dose IM.
Biological: Placebo vaccine — The placebo vaccine contains sodium chloride for injection USP, 0.9% and will be administered as a 1 mL injection IM.
  Arms: Group 3; Group 4

SUMMARY:
This study will evaluate the safety and immune response to five different combinations of three HIV vaccines in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and immune response to five different combinations of three HIV vaccines-a DNA vaccine (DNA-HIV-PT123), a NYVAC vaccine (NYVAC-HIV-PT1 and NYVAC-HIV-PT4 injections), and the AIDSVAX® B/E vaccine-in healthy, HIV-uninfected adult participants.

The study will enroll 180 healthy, HIV-uninfected participants aged 18 to 50 years. The participants will be randomly assigned to one of five groups. All participants will receive injections according to their assigned group schedule at study entry (Month 0) and Months 1, 3, and 6. The immune response of different prime and boost vaccine strategies will be tested in Groups 1 through 4, and the immune response of the co-administration of the DNA and AIDSVAX® B/E vaccine will be tested in Group 5. Group 1 participants will receive AIDSVAX® B/E as a prime followed by NYVAC as a boost; Group 2 participants will receive NYVAC as a prime followed by an AIDSVAX® B/E boost; Group 3 participants will receive AIDSVAX® B/E as a prime followed by a DNA boost; Group 4 participants will receive a DNA prime followed by an AIDSVAX® B/E boost; and Group 5 participants will receive both the DNA and AIDSVAX® B/E vaccines at each of the 4 vaccination visits.

Total study duration will be approximately 42 months and will involve 12 months of scheduled clinic visits at screening, study entry [Month 0], and Months 0.5, 1, 1.5, 3, 3.5, 6, 6.5, 9, and 12) followed by annual health contacts via e-mail or phone to a total of 3 years following initial study injection.

All study visits will include a physical exam, HIV risk reduction counseling, and an interview and/or questionnaire. Select study visits will include blood collection, urine collection, an electrocardiogram (ECG), and a pregnancy test for participants who were born female. For participants in Groups 1 and 2, select study visits will also include an assessment of cardiac symptoms. Participants will remain in the clinic for 30 minutes after receiving the vaccines for observation and monitoring. For 7 days after receiving the vaccines, participants will record their symptoms and report them to study researchers.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: participant demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years following initial study injection
* Agrees not to enroll in another study of an investigational research agent before the last required protocol clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Assessed by the clinic staff as being at "low risk" for HIV infection
* Hemoglobin greater than or equal to 11.0 g/dL for participants who were born female, greater than or equal to 13.0 g/dL for volunteers who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3
* Chemistry panel: alanine aminotransferase (ALT) less than 1.25 times the institutional upper limit of normal (IULN) and creatinine less than or equal to IULN.
* Negative HIV-1 and -2 blood test: U.S. participants must have a negative FDA-approved enzyme immunoassay (EIA). Non-U.S. sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus (anti-HCV) antibodies (Abs), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine: negative urine glucose, negative or trace urine protein, and negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range)
* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
* A participant who was born female must: agree to consistently use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. (More information on this criterion can be found in the protocol); OR not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation; OR be sexually abstinent.
* Participants who were born female must also agree not to seek pregnancy through alternative methods such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit.

Exclusion Criteria:

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45 years, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, or known hyperlipidemia
* Intent to participate in another study of an investigational research agent before the last required protocol clinic visit
* Pregnant or breastfeeding
* HIV vaccine(s) received in a prior HIV vaccine trial. For participants who have received control/placebo in an HIV vaccine trial, the HVTN 102 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For participants who have received control/placebo in an experimental vaccine trial, the HVTN 102 PSRT will determine eligibility on a case-by-case basis. For participants who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 102 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses less than 2 mg/kg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease (Not excluded: mild, well-controlled psoriasis)
* Immunodeficiency
* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the protocol.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild or moderate, well-controlled asthma. More information on this criterion can be found in the protocol.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension: If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these participants, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment. If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up)
* ECG with clinically significant findings, or features that would interfere with the assessment of myo/pericarditis, as determined by the contract ECG Lab, cardiologist, or study clinician. More information on this criterion can be found in the protocol.
* Participants who have 2 or more of the following cardiac risk factors: (1) participant report of history of elevated blood cholesterol defined as fasting low-density lipoprotein (LDL) greater than 160 mg/dL; (2) first degree relative (e.g., mother, father, brother, or sister) who had coronary artery disease before the age of 50 years); (3) current smoker; or (4) BMI greater than or equal to 35
* Allergy to eggs or egg products
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded: Participant who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure. or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if participant has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Local and systemic reactogenicity signs and symptoms | Measured up to 7 days post the last vaccination
Laboratory measures of safety | Measured through participants' last study visit at Month 12
Adverse events (AEs) and serious adverse events (SAEs) | Measured through last annual health contact at Month 36
HIV-specific binding antibody (Ab) response as assessed by binding Ab multiplex assay | Measured 2 weeks after the 4th vaccination (Month 6)
Response rate and magnitude of CD4 and CD8 T-cell responses as assessed by intracellular cytokine staining (ICS) assays | Measured 2 weeks after the 4th vaccination (Month 6)

SECONDARY OUTCOMES:
HIV-specific binding Ab and T-cell responses | Measured 2 weeks after the 4th vaccination (Month 6)
Neutralizing antibody (nAb) magnitude and breadth against tier 1 and tier 2 HIV-1 isolates as assessed by area under the magnitude-breadth curves | Measured 2 weeks after the 4th vaccination (Month 6)
HIV-specific Ab and T-cell responses | Measured 6 months after the 4th vaccination (Month 12)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Keefer, Study Chair — University of Rochester